CLINICAL TRIAL: NCT05981443
Title: Scar Analysis in Direct Excision Brow Lift: Comparing Octyl-2- Cyanoacrylate (Dermabond) Versus Non-absorbable Sutures
Brief Title: An Analysis of Dermabond vs. Non-Absorbable Sutures in Skin Closure for Brow Ptosis Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cody Blanchard (Other)
Responsible Party: Sponsor-Investigator, Cody Blanchard, Resident Physician, Ophthalmology, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BrowPtosis
Record Dates: First submitted 2023-07-31; First posted 2023-08-08 (Actual); Results first posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Brow Ptosis; Surgical Wound
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active Comparator: Dermabond (Experimental): The surgical wound over one eyebrow will be closed with Dermabond.
  Interventions: Device: Dermabond
- Active Comparator: Non-Absorbable Sutures (Active Comparator): The surgical wound over one eyebrow will be closed with non-absorbable sutures.
  Interventions: Other: Non-Absorbable Sutures

INTERVENTIONS:
Device: Dermabond — Use of Dermabond to close surgical incisions instead of non-absorbable sutures
  Arms: Active Comparator: Dermabond
Other: Non-Absorbable Sutures — Use of conventional non-absorbable sutures to close surgical incisions
  Arms: Active Comparator: Non-Absorbable Sutures

SUMMARY:
The goal of this clinical trial is to compare Dermabond with non-absorbable sutures in skin closure after brow ptosis surgery. The main questions it aims to answer are:

* if Dermabond provides equivalent wound healing compared to conventional non-absorbable skin suture techniques
* if Dermabond provides equivalent scar appearance compared to conventional non-absorbable suture techniques
* if Dermabond results in equivalent complication rates compared to conventional non-absorbable suture techniques Participants will have be randomly selected to have either Dermabond or non-absorbable suture closure methods. Scar analysis and both participant and provider surveys will be performed to assess the differences between groups, if any.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing bilateral direct excision brow lift for brow ptosis at the University of Kentucky Medical Center.
* Patients > 18 years of age.
* Patients must be able to follow up at the specified intervals.
* Patients who are able to give their own informed consent.
* Health Status: Variable health status reflective of general population of Kentucky. Patients will be healthy enough to be seen in an office setting.
* All patients will need to be proficient in the English language to understand the scale used for scar assessment

Exclusion Criteria:

* Patients <18 years of age or >100
* Allergy to Dermabond
* Adults with impaired consent capacity
* Incarcerated individuals

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Timoney, MD, Study Director — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Comparator: Dermabond | Active Comparator: Non-Absorbable Sutures
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Comparator: Dermabond | Active Comparator: Non-Absorbable Sutures | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (2) | 77 (3.7) | 73 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Scar Appearance
Description: Patient and Observer Scar Assessment Scale filled out by both patient and provider at both postoperative visits of both Dermabond and non-absorbable sutures. This survey is scaled from 0-10, with 0 being normal skin and 10 being very different skin. Lower scores are desired on this survey.
Time Frame: 10 days
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Active Comparator: Dermabond | Active Comparator: Non-Absorbable Sutures
Number analyzed (Participants) | 3 | 3
score on a scale | 7 [5 to 9] | 2.33 [1 to 4]

2. Primary Outcome: Scar Appearance
Description: as for outcome 1
Time Frame: 6 weeks
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Active Comparator: Dermabond | Active Comparator: Non-Absorbable Sutures
Number analyzed (Participants) | 3 | 3
score on a scale | 2 [1 to 3] | 4 [3 to 5]

3. Primary Outcome: Number of Participants With Complications
Description: Complications of both Dermabond and non-absorbable sutures to include dehiscence and infection
Time Frame: 6 weeks
Measure: Number; unit: participants
Arm/Group | Active Comparator: Dermabond | Active Comparator: Non-Absorbable Sutures
Number analyzed (Participants) | 3 | 3
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Active Comparator: Dermabond | Active Comparator: Non-Absorbable Sutures
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-03-30): https://cdn.clinicaltrials.gov/large-docs/43/NCT05981443/Prot_SAP_ICF_000.pdf